CLINICAL TRIAL: NCT03519997
Title: A Phase II Study of Pembrolizumab and Bavituximab in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Pembrolizumab and Bavituximab in Patients With Advanced Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Hsieh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, David Hsieh, ASSISTANT PROFESSOR- Internal Medicine - IM-Hem Onc, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102017-015
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab; bavituximab

STUDY DESIGN:
Intervention Model Description: Locally advanced or metastatic HCC not amenable to locoregional therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembro + Bavi (Experimental): Pembrolizumab 200 mg IV every 3 weeks plus, Bavituximab 3mg/kg IV weekly
  Interventions: Drug: Pembrolizumab; Drug: Bavituximab

INTERVENTIONS:
Drug: Pembrolizumab — Pembroluzumab 200mg IV once every 3 weeks
Drug: Bavituximab — Bavituximab 3mg/kg IV weekly

SUMMARY:
This is a non-randomized, open-label, multi-site phase II therapeutic trial of pembrolizumab and bavituximab in patients with locally advanced HCC. Locally advanced or metastatic HCC is defined as disease that is not amenable to surgical and/or locoregional therapies. Subjects must not have received prior systemic therapy for advanced HCC in keeping with the first-line setting of this study.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, multi-site phase II therapeutic trial of pembrolizumab and bavituximab in patients with locally advanced HCC. Locally advanced or metastatic HCC is defined as disease that is not amenable to surgical and/or locoregional therapies. Subjects must not have received prior systemic therapy for advanced HCC in keeping with the first-line setting of this study. Overall response rate (ORR) as assessed by the investigators and using RECIST 1.1 criteria, will be the primary endpoint.

Prior to initiation on treatment, all patients will sign an informed consent form. Only patients with histological proved HCC will be eligible for treatment. Tissue, either from archival formalin fixed paraffin embedded samples or a new biopsy of a target lesion will be needed.

Study therapy is defined as treatment with both pembrolizumab and bavituximab. Patients will receive trial treatment until disease progression, unacceptable toxicity, death or discontinuation from the study treatment for any other reason. Subjects will be allowed to continue study therapy after an initial investigator-assessed RECIST 1.1 defined progression as long as they meet the following criteria: 1) investigator assessed clinical benefit and 2) subject is tolerating study therapy. Subjects will be discontinued from study therapy upon the evidence of further progression, defined as an additional 10% or greater increase in tumor burden from time of initial progression (including all target lesions and new measurable lesions). New lesions are considered measurable if the longest diameter is at least 10 mm (except for pathological lymph nodes, which must have a short axis of at least 15 mm). Any new lesion considered non-measurable may become measurable and therefore included in the tumor burden measurement if the longest diameter increases to at least 10 mm (except for pathological lymph nodes, which must have an increase in short axis to at least 15 mm. For statistical analyses that include the investigator-assessed progression date, subjects who continue treatment beyond initial investigator-assessed, RECIST 1.1-defined progression will be considered to have investigator-assessed progressive disease at the time of the initial progressive event irrespective of confirmation on subsequent imaging. Patients will be followed for survival regardless of treatment discontinuation for any reason, unless they withdraw their consent to be followed for survival.

Treatment Phase

The treatment phase for each patient will begin on the initiation of study drug on Cycle 1 Day 1 (C1D1). Patients will continue study treatment until disease progression (or until discontinuation of study therapy in patient receiving pembrolizumab and bavituximab beyond progression), discontinuation due to toxicity, withdrawal of consent, or the study ends. A safety follow-up is mandatory at 30 days post the last dose.

Efficacy, safety, and correlative assessments will be performed as outlined in the Schedule of Visits and Procedures (section 6.0). Safety assessments will include hematology, biochemistry, and thyroid tests as well as ongoing evaluations of adverse events. Tumor response will be assessed radiographically every 9 weeks for the first 54 weeks, then every 12 weeks thereafter until disease progression (or until discontinuation of study therapy in patients receiving pembrolizumab or bavituximab beyond progression), loss to follow-up, or withdrawal of consent. Patients with radiological progression using RECIST may continue on study treatment if in the investigator's assessment the patient is experiencing clinical benefit and tolerating the treatment.

Dose Limiting Toxicity:

Initially, enrollment will be limited to 10 patients with no more than two patients enrolled per week. A safety committee comprised of the investigators and institutional GI Disease Orientated Team will monitor the occurrence of dose limiting toxicities (DLTs) for the first 10 patients prior to enrolling the remainder of the trial. The period for evaluating DLTs will be from the time of the first administration of study treatment through Study Day 28. DLTs will follow the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

If three or more DLTs occur during this period, enrollment will be suspended and the safety committee will make a determination of whether to reduce the bavituximab dose to 1 mg/kg. After the DLT safety assessment period for the initial 10 patients, enrollment may proceed for the remainder of the trial provided at least one patient has either a complete or partial response by RECIST 1.1 and patient safety will be evaluated on a regular basis by the institutional data safety monitoring committee (DSMC). A DLT will be defined as any treatment related toxicity in the list below that occurs during the DLT evaluation period. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded from this definition. The following will be considered DLTs:

* Any grade 4 immune-related adverse events (irAE)
* Any ≥ grade 3 colitis
* Any grade 3 or 4 noninfectious pneumonitis irrespective of duration
* Any grade 2 pneumonitis that does not resolve to grade 1 within 5 days of the initiation of maximum supportive care
* Any grade 3 irAE, excluding colitis or pneumonitis, that does not downgrade to grade 2 within 5 days of the event despite optimal medical management including systemic corticosteroids or does not downgrade to grade 1 or baseline within 14 days
* Liver transaminase elevation >8 x ULN or total bilirubin > 5 x ULN
* Any ≥ grade 3 non-irAE, except for the exclusions listed below

The definition excludes the following conditions:

* Grade 3 fatigue ≤ 7days
* Grade 3 endocrine disorder (thyroid, pituitary, and/or adrenal insufficiency) that is managed with or without systemic corticosteroid therapy and/or hormone replacement therapy and the patient is asymptomatic
* Grade 3 inflammatory reaction attributed to a local antitumor response
* Concurrent vitiligo or alopecia of any grade
* Grade 3 infusion-related reaction (first occurrence and in the absence of steroid prophylaxis) that resolves within 6 hours with appropriate clinical management
* Grade 3 or 4 neutropenia that is not associated with fever or systemic infection that improves by at least 1 grade within 3 days. Grade 3 or 4 febrile neutropenia will be considered a DLT regardless of duration or reversibility
* Grade 3 or 4 lymphopenia
* Grade 3 thrombocytopenia that is not associated with clinically significant bleeding that requires medical intervention, and improves by at least 1 grade within 3 days
* Isolated grade 3 electrolyte abnormalities that are not associated with clinical signs or symptoms and are reversed with appropriate maximal medical intervention within 3 days
* Isolated grade 3 amylase or lipase abnormalities that are not associated with clinical signs/symptoms or findings on imaging consistent with pancreatitis.

Survival follow-up phase

Patients who are no longer receiving any study treatments and have experienced disease progression will enter survival follow-up, regardless of whether they have initiated subsequent anticancer therapy. Survival follow-up information (by chart review, phone call or clinic visits) will be collected approximately every 3 months until death, loss to follow-up, withdrawal of consent or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed diagnosis hepatocellular carcinoma; known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC will be excluded
* Locally advanced or metastatic disease
* Patients with locally advanced or metastatic disease must have disease deemed not amenable to surgical and/or locoregional therapies or patients who have progressed following surgical and/or locoregional therapies.
* Measurable disease, as defined as lesions that can accurately be measured in at least one dimension according to RECIST version 1.1 at least 1 cm with contrast enhanced dynamic imaging (magnetic resonance imaging or computed tomography).
* Child-Pugh Score A
* Age ≥ 18 years
* ECOG Performance score of 0-1
* Life expectancy greater than 6 months
* Following baseline laboratory values:

  1. Total bilirubin ≤ 2.0 mg/ml
  2. INR ≤ 1.7
  3. Hgb ≥ 8.5 g/dl
  4. AST, ALT ≤5 times ULN
  5. Platelet count ≥ 50,000/mm3
  6. Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
  7. Albumin ≥ 2.5 g/dl
  8. Absolute neutrophil ≥ 1,500 cells/mm3
* Male and female subjects of child bearing potential must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
* Women of childbearing potential must have a negative pregnancy test.
* Subjects are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

HBV-HCC: Controlled (treated) hepatitis B subjects will be allowed if they meet the following criteria:

Antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Subjects on active HBV therapy with viral loads under 100 IU/ml should stay on the same therapy throughout study treatment.

Subjects who are anti-HBc (+), negative for HBsAg, negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis.

HCV-HCC: active or resolved HCV infection as evidenced by detectable HCV RNA or antibody. Patients who have failed HCV therapy as evidenced by detectable HCV RNA will be eligible. Subjects with chronic infection by HCV who are treated (successfully or treatment failure) or untreated are allowed on study. In addition, subjects with successful HCV treatment are allowed as long as there are ≥4 weeks between completion of HCV therapy and start of study drug.

Successful HCV treatment definition: SVR12.

- Prior therapy is allowed provided the following are met: at least 4 weeks since prior locoregional therapy including surgical resection, chemoembolization, radiotherapy, or ablation. Provided target lesion has increased in size by 25% or more or the target lesion was not treated with locoregional therapy. Patients treated with palliative radiotherapy for symptoms will be eligible 1 week after treatment as long as the target lesion is not the treated lesion.

Exclusion Criteria:

* Prior liver transplant;
* Patient who has received previous systemic therapy for HCC;
* Clinically significant, uncontrolled heart disease and/or recent events including any of the following:
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening;
* History of documented congestive heart failure (New York Heart Association functional classification III-IV);
* Documented cardiomyopathy;
* Patient has a left ventricular ejection fraction <40% as determined by MUGA scan or ECHO (MUGA and ECHO are not required prior to enrollment);
* Known human immunodeficiency virus (HIV) positive (testing not required);
* History of thromboembolic events (including both pulmonary embolism and deep venous thrombus but not including tumor thrombus) within the last 6 months;
* Hypersensitivity to IV contrast; not suitable for pre-medication;
* Active or fungal infections requiring systemic treatment within 7 days prior to screening;
* Known history of, or any evidence of, interstitial lung disease or active non-infectious pneumonitis;
* Evidence of poorly controlled hypertension which is defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management;
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication;
* Active, known, or suspected autoimmune disease with the following exceptions i) Subjects with vitiligo, type I diabetes mellitus, resolved childhood asthma or atopy are permitted to enroll; ii) Subjects with suspected autoimmune thyroid disorders may be enrolled if they are currently euthyroid or with residual hypothyroidism requiring only hormone replacement.

iii) Subjects with psoriasis requiring systemic therapy must be excluded from enrollment

* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the study or compromise compliance with the protocol (e.g. chronic pancreatitis, active untreated or uncontrolled fungal, bacterial, or viral infections, etc.);
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the study or compromise compliance with the protocol (e.g. chronic pancreatitis, active untreated or uncontrolled fungal, bacterial, or viral infections, etc.);
* Known history of active bacillus tuberculosis;
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days of study administration. Inhaled or topical steroids and adrenal replacement doses >10 mg/day prednisone equivalents are permitted in the absence of autoimmune disease;
* Patient who has received radiotherapy ≤ 4 weeks prior to study entry. Palliative radiotherapy for symptomatic control is acceptable (if completed at least 2 weeks prior to study drug administration and no additional radiotherapy for the same lesion is planned);
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery);
* Clinically apparent ascites on physical examination, ascites present on imaging studies is allowed;
* Patient has a known hypersensitivity to any of the excipients of bavituximab or pembrolizumab or monoclonal antibody;
* Active gastrointestinal bleeding within previous 2 months;
* History of any condition requiring anti-platelet therapy (aspirin >300 mg/day, clopidogrel >75 mg/day);
* Prisoners or subjects who are involuntarily incarcerated;
* Symptomatic or clinically active brain metastases;
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after contraception and until the termination of gestation, confirmed by a positive hCG laboratory test;
* Prior immunotherapy including anti-PD-1, anti-PD-L1, or anti-PD-L2 agents;
* Has dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and HCV infection (anti-HCV Ab(+) and detectable HCV RNA) at study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Hsieh, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health & Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembro + Bavi
Started | 35
Completed | 28
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembro + Bavi
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate (ORR) defined as the number of complete or partial responses according to RECIST 1.1 divided by the number of evaluable patients treated with combination pembrolizumab and bavituximab in patients with advanced HCC.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembro + Bavi
Number analyzed (Participants) | 28
Participants | 9

2. Secondary Outcome: Overall Survival
Description: To determine overall survival, 6-month progression free survival, and duration of response of combination pembrolizumab and bavituximab compared to historical controls
Time Frame: 36 months
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Number of Adverse Events According to the CTCAE
Description: To determine the safety and tolerability of combination pembrolizumab and bavituximab as measured by the number of adverse events according to the CTCAE 5.0
Time Frame: 36 months
Population: All patients who received at least one dose of study treatment
Measure: Number; unit: Adverse events
Arm/Group | Pembro + Bavi
Number analyzed (Participants) | 35
Adverse events | 33

ADVERSE EVENTS:
Time Frame: The planned follow-up period was 36 months. However, due to patient deaths or lost to follow-up, not all patients had follow-up data for 36 months. The actual median follow-up time was 24 months.
Description: AEs determined according to CTCAE
Arm/Group | Pembro + Bavi
All-Cause Mortality (participants affected / at risk) | 14/35
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Bavi (N=35)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
colitis (Gastrointestinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fever (Infections and infestations) | 1 (1)
acute kidney insufficiency (Renal and urinary disorders) | 2 (2)
hypoglycemia (Endocrine disorders) | 1 (1)
hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
weakness (General disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembro + Bavi (N=35)
Diarrhea (Gastrointestinal disorders) | 10
rash (Skin and subcutaneous tissue disorders) | 10
ALT increase (Hepatobiliary disorders) | 4
AST increase (Hepatobiliary disorders) | 10
Chills (General disorders) | 4
fatigue (General disorders) | 16
Neutrophil decrease (Blood and lymphatic system disorders) | 7
anemia (Blood and lymphatic system disorders) | 4
constipation (Gastrointestinal disorders) | 4
dizziness (Nervous system disorders) | 4
vomiting (Gastrointestinal disorders) | 4
fever (General disorders) | 4
headache (Nervous system disorders) | 4
anorexia (Gastrointestinal disorders) | 3
hypoglycemia (Endocrine disorders) | 3
creatinine increase (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03519997/Prot_SAP_000.pdf